CLINICAL TRIAL: NCT02283489
Title: Recombinant Human Endostatin Adenovirus Combined With Chemotherapy for Advanced Head and Neck Malignant Tumors: Phase II, Multicenter, Randomized, Controlled Clinical Trial
Brief Title: Recombinant Human Endostatin Adenovirus Combined With Chemotherapy for Advanced Head and Neck Malignant Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renmiao Zhang (Industry)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor-Investigator, Renmiao Zhang, Project leader, Chengdu Shi Endor Biological Engineering Technology Co., Ltd
Organization: Chengdu Shi Endor Biological Engineering Technology Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChengduShiEn_RMZ_001
Record Dates: First submitted 2014-10-15; First posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Head and Neck Neoplasms
Keywords: Recombinant Human Endostatin Adenovirus; Head and Neck Malignant Tumor; clinical trial; randomized; Endostatin; gene therapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Combination therapy A (Experimental): Recombinant human endostatin adenovirus (EDS01), 5.0 × 1011 VP intratumorally on days 0 and 7; paclitaxel, 160 mg/m2 intravenously on day 1; cisplatin, 25 mg/m2 intravenously on days 1 to 3.
  Interventions: Drug: recombinant human endostatin adenovirus; Drug: Cisplatin injection; Drug: Paclitaxel injection
- Combination therapy B (Experimental): Recombinant human endostatin adenovirus (EDS01), 1.0 × 1012 VP intratumorally on days 0 and 7; paclitaxel, 160 mg/m2 intravenously on day 1; cisplatin, 25 mg/m2 intravenously on days 1 to 3.
  Interventions: Drug: recombinant human endostatin adenovirus; Drug: Cisplatin injection; Drug: Paclitaxel injection
- Chemotherapy (Experimental): Paclitaxel, 160 mg/m2 intravenously on day 1; cisplatin, 25 mg/m2 intravenously on days 1 to 3.
  Interventions: Drug: Cisplatin injection; Drug: Paclitaxel injection

INTERVENTIONS:
Drug: recombinant human endostatin adenovirus — Specification: 1mL/division, 1.0×1012 virus particle (VP). ESD01 preparation: Thaw at room temperature, dilute with normal saline to required volume (no more than 2 mL).
  Method of administration: Intratumor injection, once a week for 2 weeks, every 3 weeks for one cycle. Select only one target lesion even when lesions are present. The target lesion is the largest and easiest to inject. This will be fixed during the study.
  Other Names: EDS01 (20140303)
  Arms: Combination therapy A; Combination therapy B
Drug: Cisplatin injection — Specification: 2ml: 10mg. Usage: 25mg/m2, days 1 to 3, according to instruction.
Drug: Paclitaxel injection — Specification: 5ml: 30mg. Usage: 160mg/m2 intravenously on day 1, according to instruction.

SUMMARY:
This study will investigate the efficacy and safety of recombinant human endostatin adenovirus combined with chemotherapy for advanced head and neck malignant tumors.

DETAILED DESCRIPTION:
Head and neck cancer is one of the most common malignant tumors in China, accounting for 19.9% to 30.2% of malignant tumors in this country. Approximately 60% to 70% of patients have stage III or IV disease at the time of diagnosis, and the 5-year overall survival is about 30%. The local recurrence rate ranges from 50% to 60%. The 5-year overall survival for patients treated with multidisciplinary treatment, which is a common treatment method that includes surgery, chemotherapy, radiotherapy, and biotherapy, has recently increased by 5%. Further improvements in the treatment effects of head and neck cancer are required.

Endostatin, an endogenous angiogenesis inhibitor and a C-terminal fragment of collagen XVIII, effectively inhibits tumor angiogenesis by specific inhibition of neovascular endothelial cells [7, 8]. Its characteristic antitumor effect is dose-dependent, requiring continuous high protein activity. Transportation of recombinant genes with adenovirus vectors into the body leads to continuous expression of high levels of endogenous secretory proteins, resolving the limitation of foreign protein infusion. Previous studies have shown that the antitumor activity of recombinant human endostatin adenovirus is higher than that of recombinant human endostatin protein.

EDS01, an antitumor gene therapy product that uses recombined adenovirus type 5 as the vector for the human endostatin gene, may be termed a recombinant adenovirus-recombined human endostatin gene. Intratumor injection of EDS01 reportedly results in transportation of the human endostatin gene into tumor cells by adenovirus infection, leading to the expression of endostatin protein. Expression of this protein inhibits neovascular endothelial cells, neovascularization, and tumor growth and metastasis. Both in vivo and in vitro experiments have shown that EDS01 significantly inhibits the growth of neovascular endothelial cells and tumor growth in nude mouse xenograft models of laryngocarcinoma and nasopharyngeal carcinoma.

A phase I clinical trial (No. treatment effect) conducted at West China Hospital of Sichuan University enrolled patients with superficial advanced head and neck cancer lesions. The patients underwent injection of different doses of EDS01, and the investigators performed a preliminary evaluation of the maximally tolerated dose and adverse events. The study showed that, whether administered by dose escalation or in multiple doses, EDS01 was well tolerated without dose-limiting toxicity and maximum tolerated dose. The main side effects were fever and injection site pain with flu-like symptoms. A small amount of EDS01 (1/10 000 000) was absorbed into the bloodstream. A thimbleful (1/100 000 000 to 1/10 000 000 000) was excreted in the urine and feces and was nontoxic to the environment. The target lesions exhibited a treatment response.

According to the results of this phase I trial, both 5.0 × 1011 and 1.0 × 1012 virus particles (VP) of EDS01 showed adequate safety and treatment responses. Therefore, in the subsequent phase II clinical trial, the optimal of these two doses will be determined. The treatment effects and safety of this protocol for head and neck cancer will also be further investigated.

In summary, this study will initially explore the efficacy and safety of recombinant human endostatin adenovirus combined with chemotherapy for advanced head and neck malignant tumors.

In the experimental group, the target lesion is defined as that injected by EDS01. In the control group, the target lesion is defined as that selected at the inception.

ELIGIBILITY:
Inclusion Criteria:

* Advanced head and neck cancer unsuitable for surgery or radiotherapy (including head and neck squamous carcinoma and nasopharyngeal carcinoma, which should not more than 30%)
* Cytological and/or histopathologic diagnosis
* Target lesions can be treated with intratumor injection
* Lesions can be measured by imaging with a diameter of ≥2 cm (RECIST1.1)
* No chemotherapy, radiotherapy, or biotherapy administered in the past 4 weeks
* Age of 18 to 70 years
* Life expectation of ≥12 weeks
* ECOG performance status of 0 to 2
* Laboratory examinations performed ≤7 days before enrollment with the following results: absolute neutrophil count of ≥1.5 × 109 L-1, platelet count of ≥80 × 109/L, total bilirubin level of ≤2 mg/dL, AST and ALT levels of ≤2 times the upper limit of the reference range, and coagulation parameters ≤1.5 times the upper limit of the reference range
* Voluntary participation and written informed consent

Exclusion Criteria:

* Allergy to EDS01
* Nerves and vessels passing through target lesions do not allow for injection of EDS01 into lesions
* Simultaneous radiation of target lesions
* Cancer recurrence within 6 months treated by paclitaxel
* Severe coagulation dysfunction and bleeding tendency
* Serious medical diseases, myocardial infraction in the past 3 months, or acute infection
* Currently pregnant or lactating
* Any conditions that the investigator regards as unsuitable for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Change in Objective response rate (ORR) of target lesion | During the 2nd and 4th cycle of treatment phase (day 35, day 76) and follow-up (every 3 months after treatment till 2 years).
  Objective response rate (ORR) of target lesion is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR), , determined by tumor assessments from radiological tests including CT and MRI. CR is defined as disappearance of the target lesion. PR is defined as a decrease of at least 30% in the product of two perpendicular diameters of the target lesion.

SECONDARY OUTCOMES:
Change in Disease control rate of target lesion | During the 2nd and 4th cycle of treatment phase (day 35, day 76) and follow-up (every 3 months after treatment till 2 years).
  The disease control rate of the target lesion includes CR, PR, and stable disease (SD). SD is defined as a decrease of <30% or an increase of <20% in the size of the target lesion, determined by tumor assessments from radiological tests including CT and MRI.
Change in ORR of all lesions | During the 2nd and 4th cycle of treatment phase (day 35, day 76) and follow-up (every 3 months after treatment till 2 years).
  All lesions include the target lesions, nontarget lesions, and new lesions. ORR of all lesions includes CR and PR.
Time to progression | Up to 24 weeks
  Time to progression is defined as the time from randomization until objective tumor progression as verified for the first time.
Change in Immune response | During the screening phase and on days 7, 21, 35, 48, 62, and 76 (day 1 is defined as the first day of chemotherapy with the TP regimen)
  Serum IgG antibody responses to the respective viruses will be detected in blood samples. ELISA will be used to test the quantity of serum IgG in a central laboratory according to the specific provisions of the central laboratory. During the screening phase and on days 7, 21, 35, 48, 62, and 76, venous serum (3 mL) will be gathered in a drying tube by venipuncture. After 30 minutes, they will be centrifuged at 2 000 r/min for 10 minutes, and the supernatant will be stored at -80 °C for testing.

OTHER OUTCOMES:
Change in adenovirus in patients' secreta and excreta | Before the first administration and on days 1 and 3 after the first administration
  Only the leading center will be tested for environmental pollution. This testing will include evaluation of swab specimens, urine specimens, and fecal specimens before the first administration and immediately, 24 hours, and 3 days after the first administration. Specimens will be taken from injection sites and the oropharynx and stored at -80 °C for testing. Urine specimens (2 mL) will be gathered at different times and mixed, then stored at -80 °C for testing. Feces will be gathered in tubes, mixed with 2 mL of normal saline, stirred for 5 minutes, and centrifuged at 2 000 r/min for 10 minutes; the supernatant will be stored at -80 °C for testing.
Change in vital signs and physique | Screening phase (before randomization) and treatment phase (until week 12 after treatment)
  Laboratory examination: complete blood count, routine urinalysis, routine fecal test, liver function, renal function, and electrolytes. Coagulation tests will be performed on the first day of the first cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Renmiao Zhang, MD, PhD, Study Director — Chengdu Shi Endor Biological Engineering Technology Co., Ltd
Locations (4):
- China (4):
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Chongqing Cancer Hospital, Chongqing
  - Shanghai Ninth People's Hospital Affiliated Shanghai JiaoTong University School of Medicine, Shanghai